CLINICAL TRIAL: NCT01796470
Title: A Phase 2, Open-Label Study Evaluating the Efficacy, Safety, Tolerability, and Pharmacodynamics of GS-9973 in Combination With Idelalisib in Subjects With Relapsed or Refractory Hematologic Malignancies
Brief Title: Entospletinib in Combination With Idelalisib in Adults With Relapsed or Refractory Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to safety measures.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-339-0103
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma; Diffuse Large B-cell Lymphoma; Indolent Non-Hodgkin's Lymphoma
Keywords: GS-US-339-0103; SYK inhibitor; PI3K inhibitor; GS-9973; GS 9973; GS-1101; GS 1101; Cal-101; Cal 101; idelalisib; leukemia; lymphoma; CLL; MCL; DLBCL; iNHL; FL; MZL; LPL; SLL; WM; Waldenström's macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Leukemia; Lymphoma; Waldenstrom Macroglobulinemia | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entospletinib + idelalisib (Experimental): Entospletinib plus idelalisib at one of 4 dose combinations (400 mg/100 mg; 600 mg/100 mg; 800 mg/100 mg; 800 mg/150 mg).
  After discontinuation of entospletinib+idelalisib combination therapy, and following a washout period, participants may continue to receive entospletinib 400 mg monotherapy.
  Interventions: Drug: Entospletinib; Drug: Idelalisib

INTERVENTIONS:
Drug: Entospletinib — Entospletinib tablets administered orally twice daily
  Other Names: GS-9973
Drug: Idelalisib — Idelalisib tablets administered orally twice daily
  Other Names: GS-1101; GS 1101; Cal-101; Cal 101; Zydelig®

SUMMARY:
This study will evaluate the efficacy of the combination entospletinib and idelalisib in participants with relapsed or refractory hematologic malignancies. Participants will be enrolled who have one of the following hematological tumor types: chronic lymphocytic leukemia (CLL), mantle cell lymphoma (MCL), diffuse large B-cell lymphoma (DLBCL), or indolent non-Hodgkin lymphomas (iNHL; including follicular lymphoma (FL) and lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia [LPL/WM], small lymphocytic lymphoma [SLL], or marginal zone lymphoma [MZL]).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of B-cell indolent non-Hodgkin lymphoma (iNHL),diffuse large B-cell lymphoma (DLBCL),mantle cell lymphoma (MCL), or chronic lymphocytic leukemia (CLL) as documented by medical records and with histology based on criteria established by the World Health Organization
* For institutions that have Phase 3 or Phase 4 protocols studying idelalisib (Zydelig®; GS-1101); individuals with malignancies being studied in these protocols must have failed screening and be registered as a screen failure in the respective idelalisib protocol
* Prior treatment for lymphoid malignancy
* Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy
* Discontinuation of all therapy for the treatment of cancer ≥ 3 weeks before the start of study drug
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤ 1 before the start of study drug
* Karnofsky performance status of ≥ 60
* Life expectancy of at least 3 months

Key Exclusion Criteria:

* Known histological transformation from iNHL or CLL to an aggressive form of NHL (ie, Richter transformation)
* Known active central nervous system or leptomeningeal lymphoma
* Presence of known intermediate- or high-grade myelodysplastic syndrome
* Current therapy with agents that reduce gastric acidity, including but not limited to antacids, H2 inhibitors, and proton pump inhibitors
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of start of study drug
* Ongoing liver injury
* Ongoing or recent hepatic encephalopathy
* Ongoing drug-induced pneumonitis
* Ongoing inflammatory bowel disease
* Ongoing alcohol or drug addiction
* Pregnancy or breastfeeding
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy
* Concurrent participation in an investigational drug trial with therapeutic intent

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- United States (13):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Collaborative Research Group LLC, Boynton Beach, Florida
  - Weill Cornell Medical College, New York, New York
  - University of Rochester, James P. Wilmot Cancer Center, Rochester, New York
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Charleston Hematology Oncology, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties, Tacoma, Washington

REFERENCES:
- [Derived] Barr PM, Saylors GB, Spurgeon SE, Cheson BD, Greenwald DR, O'Brien SM, Liem AK, Mclntyre RE, Joshi A, Abella-Dominicis E, Hawkins MJ, Reddy A, Di Paolo J, Lee H, He J, Hu J, Dreiling LK, Friedberg JW. Phase 2 study of idelalisib and entospletinib: pneumonitis limits combination therapy in relapsed refractory CLL and NHL. Blood. 2016 May 19;127(20):2411-5. doi: 10.1182/blood-2015-12-683516. Epub 2016 Mar 11. PMID 26968534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 20 June 2013. The last study visit occurred on 22 December 2016.
Pre-assignment Details: 85 participants were screened.
Groups:
- Entospletinib + Idelalisib CLL: Participants with a documented diagnosis of chronic lymphocytic leukemia (CLL) were included in this arm. Participants were administered 4 dose combinations of entospletinib plus idelalisib tablets orally twice daily under fasted conditions (400 mg/100 mg for 2 weeks, if no dose limiting toxicity (DLT) occurred, increased dose to 600 mg/100 mg for 2 weeks, if no DLT occurred, increased dose to 800 mg/100 mg for 4 weeks, if no DLT occurred, increased dose to 800 mg/150 mg) for up to 6 months. After discontinuation of combination therapy and a washout period of 14-28 days, participants could continue to receive entospletinib 400 mg monotherapy for up to 18 months.
- Entospletinib + Idelalisib iNHL: FL: Participants with a documented diagnosis of indolent non-Hodgkin lymphoma (iNHL) with follicular lymphoma (FL) were included in this arm. Participants were administered 4 dose combinations of entospletinib plus idelalisib tablets orally twice daily under fasted conditions (400 mg/100 mg for 2 weeks, if no dose limiting toxicity (DLT) occurred, increased dose to 600 mg/100 mg for 2 weeks, if no DLT occurred, increased dose to 800 mg/100 mg for 4 weeks, if no DLT occurred increased dose to 800 mg/150 mg) for up to 6 months. After discontinuation of combination therapy and a washout period of 14-28 days, participants could continue to receive entospletinib 400 mg monotherapy for up to 18 months.
- Entospletinib + Idelalisib DLBCL: Participants with a documented diagnosis of diffuse large B-cell lymphoma (DLBCL) were included in this arm. Participants were administered 4 dose combinations of entospletinib plus idelalisib tablets orally twice daily under fasted conditions (400 mg/100 mg for 2 weeks, if no dose limiting toxicity (DLT) occurred ,increased dose to 600 mg/100 mg for 2 weeks, if no DLT occurred, increased dose to 800 mg/100 mg for 4 weeks, if no DLT occurred, increased dose to 800 mg/150 mg) for up to 6 months. After discontinuation of combination therapy and a washout period of 14-28 days, participants could continue to receive entospletinib 400 mg monotherapy for up to 18 months.
- Entospletinib + Idelalisib MCL: Participants with a documented diagnosis of mantle cell lymphoma (MCL) were included in this arm. Participants were administered 4 dose combinations of entospletinib plus idelalisib tablets orally twice daily under fasted conditions (400 mg/100 mg for 2 weeks, if no dose limiting toxicity (DLT) occurred, increased dose to 600 mg/100 mg for 2 weeks, if no DLT occurred, increased dose to 800 mg/100 mg for 4 weeks, if no DLT occurred, increased dose to 800 mg/150 mg) for up to 6 months. After discontinuation of combination therapy and a washout period of 14-28 days, participants could continue to receive entospletinib 400 mg monotherapy for up to 18 months.
- Entospletinib + Idelalisib iNHL: Others: Participants with a documented diagnosis of iNHL with other subtypes lymphoplasmacytic lymphoma (LPL)/Waldenstrom macroglobulinemia (WM), small lymphocytic lymphoma (SLL), and marginal zone lymphoma (MZL) were included in this arm. Participants were administered 4 dose combinations of entospletinib plus idelalisib tablets orally twice daily under fasted conditions (400 mg/100 mg for 2 weeks, if no dose limiting toxicity (DLT) increased to 600 mg/100 mg for 2 weeks, if no DLT increased to 800 mg/100 mg for 4 weeks, if no DLT increased to 800 mg/150 mg) for up to 6 months. After discontinuation of combination therapy and a washout period of 14-28 days, participants could continue to receive entospletinib 400 mg monotherapy for up to 18 months.
Period: Overall Study
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Started | 35 | 14 | 6 | 3 | 8
Entospletinib Monotherapy (Participants who received monotherapy when combination therapy was discontinued.) | 4 | 4 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 35 | 14 | 6 | 3 | 8
Not completed — Adverse Event | 4 | 2 | 2 | 1 | 3
Not completed — Death | 2 | 0 | 0 | 0 | 1
Not completed — Initiated New Therapy | 9 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 5 | 4 | 1 | 0 | 1
Not completed — Progressive Disease | 7 | 7 | 3 | 2 | 0
Not completed — Protocol Criteria for Withdrawal | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set comprised all participants who received ≥ 1 dose of study drug (entospletinib or idelalisib).
Groups:
- Entospletinib + Idelalisib iNHL: Others: Participants with a documented diagnosis of iNHL with other subtypes lymphoplasmacytic lymphoma (LPL)/Waldenstrom macroglobulinemia (WM), small lymphocytic lymphoma (SLL) and marginal zone lymphoma (MZL) were included in this arm. Participants were administered 4 dose combinations of entospletinib plus idelalisib tablets orally twice daily under fasted conditions (400 mg/100 mg for 2 weeks, if no dose limiting toxicity (DLT) increased to 600 mg/100 mg for 2 weeks, if no DLT increased to 800 mg/100 mg for 4 weeks, if no DLT increased to 800 mg/150 mg) for up to 6 months. After discontinuation of combination therapy and a washout period of 14-28 days, participants could continue to receive entospletinib 400 mg monotherapy for up to 18 months.
- Total: Total of all reporting groups
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others | Total
Number analyzed (Participants) | 35 | 14 | 6 | 3 | 8 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (12.9) | 64 (13.4) | 69 (17.4) | 62 (10.8) | 69 (8.9) | 67 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 4 | 1 | 5 | 31
  Male | 20 | 8 | 2 | 2 | 3 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted Category used, as local regulators did not allow collection of race or ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Ethnicity: Not Hispanic or Latino | 35 | 12 | 6 | 3 | 8 | 64
    Ethnicity: Not Permitted | 0 | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 27 | 11 | 6 | 3 | 8 | 55
  Race: Black or African American | 5 | 1 | 0 | 0 | 0 | 6
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Race: Asian | 2 | 0 | 0 | 0 | 0 | 2
  Race: Other | 0 | 1 | 0 | 0 | 0 | 1
  Race: Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Karnofsky Performance Status [Count of Participants; unit: Participants] — Karnofsky Performance Status will be assessed on a scale of 0-100 where 0 indicates death and 100 indicates normal activity.
  Participants
    40 | 1 | 0 | 0 | 0 | 0 | 1
    50 | 1 | 0 | 0 | 0 | 0 | 1
    60 | 2 | 0 | 0 | 1 | 0 | 3
    70 | 2 | 1 | 1 | 0 | 0 | 4
    80 | 9 | 7 | 2 | 1 | 5 | 24
    90 | 14 | 4 | 3 | 1 | 3 | 25
    100 | 6 | 2 | 0 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR assessed by the Independent Review Committee (IRC), was based on the International Working Group Revised Response Criteria (Cheson, 2012) and investigator's response, defined as the percentage of participants achieving a complete response (CR) or partial response (PR) (or very good partial response [VGPR] or minor response [MR] for participants with LPL/WM). CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. PR was defined as a ≥ 50% reduction in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions. VGPR and MR were defined as ≥ 90% and ≥ 25% but < 50% decrease from baseline in serum monoclonal immunoglobulin M (IgM) concentration by serum protein electrophoresis (SPEP) respectively.
Time Frame: Start of treatment to end of treatment (Up to 18 months)
Population: The study was terminated due to safety measures. Complete data was not collected for any participant.
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Description: A treatment-emergent Adverse Event (AE) was defined as any AE with an onset date of on or after the study drug start date and no later than 30 days after permanent discontinuation of study drugs or an AE leading to premature discontinuation of study drug. An AE is any untoward medical occurrence in a clinical investigation where participants administered a medicinal product, and which does not necessarily have a causal relationship with this treatment.
Time Frame: First dose date up to the last dose date plus 30 days (maximum duration: 19 months)
Population: The Safety Analysis Set comprised all participants who received ≥ 1 dose of study drug (entospletinib or idelalisib).
Measure: Number; unit: percentage of participants
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Number analyzed (Participants) | 35 | 14 | 6 | 3 | 8
percentage of participants | 100 | 100 | 100 | 100 | 100

3. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory (Hematology, Serum Chemistry and Urinalysis) abnormality was defined as an abnormality that, compared to baseline, worsens by ≥ 1 grade in the period from the first dose of study drug. Safety as assessed by grading of laboratory values and AEs according to the National Cancer Institutes' Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. Grade 0 = none, Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening or disabling. If baseline data are missing, then any graded abnormality (i.e., an abnormality that is Grade ≥ 1 in severity) will be considered treatment-emergent. The percentage of participants in each worst postbaseline grade is reported.
Time Frame: First dose date up to the last dose date plus 30 days (maximum: 18 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Entospletinib + Idelalisib iNHL: Others: Participants with a documented diagnosis of iNHL with other subtypes lymphoplasmacytic lymphoma (LPL)/ Waldenstrom macroglobulinemia (WM), small lymphocytic lymphoma (SLL), and marginal zone lymphoma (MZL) were included in this arm. Participants were administered 4 dose combinations of entospletinib plus idelalisib tablets orally twice daily under fasted conditions (400 mg/100 mg for 2 weeks, if no dose limiting toxicity (DLT) increased to 600 mg/100 mg for 2 weeks, if no DLT increased to 800 mg/100 mg for 4 weeks, if no DLT increased to 800 mg/150 mg) for up to 6 months. After discontinuation of combination therapy and a washout period of 14-28 days, participants could continue to receive entospletinib 400 mg monotherapy for up to 18 months.
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Number analyzed (Participants) | 35 | 14 | 6 | 3 | 8
percentage of participants
  Neutrophils Count Decreased (Grade 1) | 17.1 | 21.4 | 0 | 66.7 | 25.0
  Neutrophils Count Decreased (Grade 2) | 20.0 | 14.3 | 0 | 0 | 25.0
  Neutrophils Count Decreased (Grade 3) | 14.3 | 7.1 | 16.7 | 0 | 0
  Neutrophils Count Decreased (Grade 4) | 11.4 | 7.1 | 0 | 0 | 25.0
  Anemia (Grade 1) | 20.0 | 35.7 | 16.7 | 0 | 0
  Anemia (Grade 2) | 14.3 | 7.1 | 16.7 | 0 | 0
  Anemia (Grade 3) | 5.7 | 0 | 16.7 | 0 | 0
  Anemia (Grade 4) | 0 | 0 | 0 | 0 | 0
  Leukocytosis (Grade 1) | 0 | 0 | 0 | 0 | 0
  Leukocytosis (Grade 2) | 0 | 0 | 0 | 0 | 0
  Leukocytosis (Grade 3) | 28.6 | 0 | 0 | 33.3 | 0
  Leukocytosis (Grade 4) | 0 | 0 | 0 | 0 | 0
  White Blood Cell Count Decreased (Grade 1) | 0 | 21.4 | 16.7 | 0 | 12.5
  WBC Count Decreased (Grade 2) | 14.3 | 0 | 16.7 | 33.3 | 12.5
  WBC Count Decreased (Grade 3) | 5.7 | 14.3 | 0 | 0 | 12.5
  WBC Count Decreased (Grade 4) | 0 | 0 | 0 | 0 | 12.5
  Lymphocyte Count Decreased (Grade 1) | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased (Grade 2) | 0 | 0 | 16.7 | 33.3 | 12.5
  Lymphocyte Count Decreased (Grade 3) | 5.7 | 21.4 | 50.0 | 0 | 12.5
  Lymphocyte Count Decreased (Grade 4) | 0 | 0 | 0 | 33.3 | 0
  Lymphocyte Count Increased (Grade 1) | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased (Grade 2) | 8.6 | 7.1 | 16.7 | 0 | 0
  Lymphocyte Count Increased (Grade 3) | 28.6 | 0 | 0 | 0 | 12.5
  Lymphocyte Count Increased (Grade 4) | 0 | 0 | 0 | 0 | 0
  Platelets Count Decreased (Grade 1) | 11.4 | 28.6 | 16.7 | 33.3 | 0
  Platelets Count Decreased (Grade 2) | 2.9 | 7.1 | 0 | 0 | 0
  Platelets Count Decreased (Grade 3) | 5.7 | 14.3 | 0 | 0 | 0
  Platelets Count Decreased (Grade 4) | 2.9 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT) Increased (Grade 1) | 22.9 | 7.1 | 33.3 | 0 | 50.0
  ALT Increased (Grade 2) | 8.6 | 7.1 | 0 | 0 | 0
  ALT Increased (Grade 3) | 0 | 35.7 | 16.7 | 33.3 | 0
  ALT Increased (Grade 4) | 5.7 | 0 | 0 | 0 | 12.5
  Hypoalbuminemia (Grade 1) | 14.3 | 28.6 | 0 | 0 | 12.5
  Hypoalbuminemia (Grade 2) | 5.7 | 0 | 16.7 | 33.3 | 0
  Hypoalbuminemia (Grade 3) | 0 | 0 | 16.7 | 0 | 0
  Hypoalbuminemia (Grade 4) | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (ALP) Increased (Grade 1) | 17.1 | 28.6 | 33.3 | 33.3 | 12.5
  ALP Increased (Grade 2) | 2.9 | 0 | 0 | 0 | 12.5
  ALP Increased (Grade 3) | 0 | 0 | 0 | 0 | 0
  ALP Increased (Grade 4) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST)Increased(Grade 1) | 20.0 | 14.3 | 50.0 | 0 | 37.5
  AST Increased (Grade 2) | 2.9 | 14.3 | 0 | 33.3 | 0
  AST Increased (Grade 3) | 0 | 28.6 | 16.7 | 0 | 12.5
  AST Increased (Grade 4) | 5.7 | 0 | 0 | 0 | 0
  Chronic Kidney Disease (Grade 1) | 34.3 | 42.9 | 50.0 | 33.3 | 37.5
  Chronic Kidney Disease (Grade 2) | 0 | 7.1 | 33.3 | 0 | 0
  Chronic Kidney Disease (Grade 3) | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease (Grade 4) | 0 | 0 | 0 | 0 | 0
  Hyperglycemia (Grade 1) | 11.4 | 7.1 | 0 | 0 | 12.5
  Hyperglycemia (Grade 2) | 5.7 | 7.1 | 0 | 0 | 0
  Hyperglycemia (Grade 3) | 11.4 | 0 | 0 | 0 | 0
  Hyperglycemia (Grade 4) | 0 | 0 | 0 | 0 | 0
  Hypoglycemia (Grade 1) | 0 | 14.3 | 0 | 33.3 | 25.0
  Hypoglycemia (Grade 2) | 0 | 0 | 0 | 0 | 0
  Hypoglycemia (Grade 3) | 0 | 0 | 0 | 0 | 0
  Hypoglycemia (Grade 4) | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia (Grade 1) | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia (Grade 2) | 2.9 | 7.1 | 0 | 0 | 0
  Hypophosphatemia (Grade 3) | 5.7 | 0 | 16.7 | 0 | 12.5
  Hypophosphatemia (Grade 4) | 0 | 0 | 0 | 0 | 0
  Hypokalemia (Grade 1) | 20.0 | 7.1 | 33.3 | 0 | 0
  Hypokalemia (Grade 2) | 0 | 0 | 0 | 0 | 0
  Hypokalemia (Grade 3) | 0 | 0 | 0 | 0 | 0
  Hypokalemia (Grade 4) | 0 | 0 | 0 | 0 | 0
  Hyponatremia (Grade 1) | 20.0 | 0 | 50.0 | 0 | 0
  Hyponatremia (Grade 2) | 0 | 0 | 0 | 0 | 0
  Hyponatremia (Grade 3) | 5.7 | 0 | 0 | 0 | 25.0
  Hyponatremia (Grade 4) | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased (Grade 1) | 17.1 | 14.3 | 50.0 | 0 | 12.5
  Blood Bilirubin Increased (Grade 2) | 25.7 | 14.3 | 16.7 | 0 | 0
  Blood Bilirubin Increased (Grade 3) | 2.9 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased (Grade 4) | 0 | 0 | 0 | 0 | 0
  Proteinuria (Grade 1) | 22.9 | 7.1 | 0 | 0 | 12.5
  Proteinuria (Grade 2) | 2.9 | 14.3 | 0 | 0 | 0
  Proteinuria (Grade 3) | 0 | 0 | 0 | 0 | 0
  Proteinuria (Grade 4) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Tolerated Dose Level
Description: Maximum tolerated dose (MTD) is defined as the highest dose level that was consistently well tolerated without dose limiting toxicity (DLT) for the majority of participants time on treatment (ie,> 50%) as determined by the investigator for each participant. DLTs are defined as Grade 4 hematological toxicities persisting for ≥ 14 days or Grade ≥ 3 toxicities of other types.
Time Frame: First dose (entospelinib + idelalisib) date up to 6 months
Population: The study was terminated due to safety measures. Complete data was not collected for any participant.
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval from the first dose of study drug to the earlier of the first documentation of definitive disease progression or death from any cause.
Time Frame: Start of treatment to end of treatment (Up to 18 months)
Population: The study was terminated due to safety measures. Complete data was not collected for any participant.
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the interval from the first-time response (CR or PR [or VGPR or MR for participants with LPL/WM]) is achieved to the earlier of the first documentation of definitive disease progression or death from any cause.CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. PR was defined as a ≥ 50% reduction in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions. VGPR and MR were defined as ≥ 90% and ≥ 25% but < 50% decrease from baseline in serum monoclonal IgM concentration by SPEP respectively.
Time Frame: Start of treatment to end of treatment (Up to 18 months)
Population: The study was terminated due to safety measures. Complete data was not collected for any participant.
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the interval from the first dose of entospletinib/idelalisib to the time response (CR or PR [or VGPR or MR for participants with LPL/WM]) is first achieved. CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. PR was defined as a ≥ 50% reduction in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions. VGPR and MR were defined as ≥ 90% and ≥ 25% but < 50% decrease from baseline in serum monoclonal IgM concentration by SPEP respectively.
Time Frame: Start of treatment to end of treatment (Up to 18 months)
Population: The study was terminated due to safety measures. Complete data was not collected for any participant.
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date plus 30 days (maximum duration: 19 months); All-Cause Mortality: Baseline to Last Follow-Up Visit (Up to 3.6 years)
Description: The Safety Analysis Set comprised all participants who received ≥ 1 dose of study drug (entospletinib or idelalisib).
Arm/Group | Entospletinib + Idelalisib CLL | Entospletinib + Idelalisib iNHL: FL | Entospletinib + Idelalisib DLBCL | Entospletinib + Idelalisib MCL | Entospletinib + Idelalisib iNHL: Others
All-Cause Mortality (participants affected / at risk) | 3/35 | 1/14 | 2/6 | 2/3 | 2/8
Serious Adverse Events (participants affected / at risk) | 24/35 | 2/14 | 4/6 | 2/3 | 5/8
Other Adverse Events (participants affected / at risk) | 34/35 | 14/14 | 6/6 | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entospletinib + Idelalisib CLL (N=35) | Entospletinib + Idelalisib iNHL: FL (N=14) | Entospletinib + Idelalisib DLBCL (N=6) | Entospletinib + Idelalisib MCL (N=3) | Entospletinib + Idelalisib iNHL: Others (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Drug interaction (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 5 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entospletinib + Idelalisib CLL (N=35) | Entospletinib + Idelalisib iNHL: FL (N=14) | Entospletinib + Idelalisib DLBCL (N=6) | Entospletinib + Idelalisib MCL (N=3) | Entospletinib + Idelalisib iNHL: Others (N=8)
Anaemia (Blood and lymphatic system disorders) | 5 | 0 | 2 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 11 | 2 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 2 | 2 | 0 | 1
Dyschezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 0 | 2 | 1 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 14 | 7 | 4 | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 2 | 2 | 0 | 1
Asthenia (General disorders) | 3 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 1 | 0 | 0
Chills (General disorders) | 7 | 1 | 3 | 0 | 1
Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 15 | 6 | 4 | 0 | 3
Malaise (General disorders) | 3 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 5 | 1 | 1 | 0 | 1
Pain (General disorders) | 2 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 10 | 5 | 5 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 4 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 5 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 4 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 7 | 4 | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 1 | 0 | 0
International normalised ratio abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 1 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 4 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 2 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 9 | 4 | 1 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 1 | 2 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 1 | 2 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
As a result of the early termination of the trial for safety, the efficacy endpoints were not evaluable due to insufficient treatment exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years